CLINICAL TRIAL: NCT06699381
Title: Investigation Of The Relationship Between Spinal Straightness And Posture And Balance, Physical Performance And Energy Consumption In Individuals With Stroke
Brief Title: Spinal Straightness, Posture And Balance, Physical Performance And Energy Consumption In Individuals With Stroke
Status: Recruiting | Type: Observational
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Saniye Aydoğan Arslan, assoc. prof. dr., Kırıkkale University
Other Study IDs: KirikkaleU-SCEYLAN-001
Record Dates: First submitted 2024-09-25; First posted 2024-11-21 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Stroke; Postural; Defect; Energy Supply; Deficiency
Keywords: stroke,posture,balance,spinal straightness
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stroke: Descriptive research
  Interventions: Device: use of spinal mouse; Diagnostic Test: Brunnstrom's Hemiplegia Recovery Staging; Diagnostic Test: The six minute walking test (6MWT); Diagnostic Test: Functional Reach Test (FRT); Diagnostic Test: Mini Balance Evaluation Systems Test (Mini-BESTest); Diagnostic Test: The five Times Sit to Stand Test (5x Sit-To-Stand Test); Diagnostic Test: The Postural Assessment Scale for Stroke (PASS); Diagnostic Test: Postural Symmetry Index and Weight Transfer Symmetry; Diagnostic Test: Measurement of the craniovertebral angle

INTERVENTIONS:
Device: use of spinal mouse — Spinal Mouse (SM) is an external non-invasive measurement device that evaluates the spinal angle and shape in the frontal and sagittal planes
Diagnostic Test: Brunnstrom's Hemiplegia Recovery Staging — According to Brunnstrom's stages of recovery, the individual will be identified at which stage
Diagnostic Test: The six minute walking test (6MWT) — It evaluates the functional capacity of the individual and it provides valuable information regarding all the systems during physical activity, including pulmonary and cardiovascular systems, blood circulation, neuromuscular units, body metabolism, and peripheral circulation
Diagnostic Test: Functional Reach Test (FRT) — Functional Reach Test (FRT) is a clinical outcome measure and assessment tool for ascertaining dynamic balance in in simple task.
  In standing, measures the distance between the length of an outstretched arm in a maximal forward reach, while maintaining a fixed base of support.
  This information is correlated with risk of falling A number of factors exert a major influence on this evaluation: Research revealed that movement strategy and reduced spinal flexibility both affect reach distance.
Diagnostic Test: Mini Balance Evaluation Systems Test (Mini-BESTest) — This test measures dynamic balance, functional mobility, and gait. It is commonly used in populations who have or have had multiple sclerosis (MS), Parkinson disease (PD), strokes, spinal cord injury (SCI), or cancer.
  The Mini-BESTest was developed in 2010 from the Balance Evaluation Systems Test (BESTest), then revised in 2013 to clarify inconsistencies in scoring. The scoring instructions were different in the published and online versions. The revision clarified that the Mini-BESTest should be scored out of 28 points. Explanations for how to score items 3, 6, and 14 were also given.
  The Mini-BESTest consists of 14 items, including 4 of the 6 sections (anticipatory postural adjustments, reactive postural control, sensory orientation, and dynamic gait) from the BESTest.
Diagnostic Test: The five Times Sit to Stand Test (5x Sit-To-Stand Test) — It's used to asses functional lower limbs strength, transitional movements, balance, and fall risk in older adults.
Diagnostic Test: The Postural Assessment Scale for Stroke (PASS) — The Postural Assessment Scale for Stroke (PASS) is an outcome measure specifically designed to assess and monitor postural control after stroke. It was developed in 1999 as an adaptation of the Fugl-Meyer Assessment balance subscale[1]. It contains 12 four-level items of varying difficulty for assessing ability to maintain or change a given lying, sitting or standing posture
Diagnostic Test: Postural Symmetry Index and Weight Transfer Symmetry — It is a form of measurement in which two scales are used to calculate the weight transferred to the intact and stroke limb. The values obtained as a result of the test are calculated with formulas.
Diagnostic Test: Measurement of the craniovertebral angle — Measurement of the craniovertebral angle; the patient is asked to find the most natural position by flexion and extension of the head in the standing position and a photograph is taken with a digital camera from a distance of 1.5 m to the shoulder level of the patient and this process is repeated 3 times. The images obtained are then digitally calculated with the help of an appropriate program.

SUMMARY:
Patients diagnosed with ischemic or hemorrhagic stroke who applied to Kırıkkale University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation will be included in the study. The aim of our study is to investigate the relationship between spinal alignment, posture and weight transfer symmetry with balance, physical performance and energy expenditure in stroke patients.

DETAILED DESCRIPTION:
Patients diagnosed with ischemic or hemorrhagic stroke who applied to Kırıkkale University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation will be included in the study. The number of patients to be included in our study will be determined by power analysis.

Sociodemographic information (Age, Gender, Body Mass Index, Dominant Side) of the individuals included in the study will be recorded.

Information about the stroke (cause of stroke, time elapsed since stroke, side of involvement, neglect after stroke, comorbidities, history of falls in the last six months and 1 year, use of assistive devices, etc.) will be recorded.

1. Motor assessment The motor level of the individuals will be assessed according to the Brunnstrom Assessment. Upper and lower extremities will be evaluated separately.
2. Posture assessment Within the scope of the posture assessment of the individuals, Spinal Mouse, a computer-aided device, will be used for spinal alignment, and Postural Symmetry Index and Weight Transfer Symmetry will be calculated.
3. Balance Trunk control will be assessed with the Postural Assessment Scale for Stroke Patients (PASS), standing balance will be assessed with the Minibestest, Functional reach test (FUT) and timed get up and walk test (ZKTY)
4. Physical performance assessment Six-minute walk test and 5 times sit and stand test will be used to evaluate physical performance. In addition, physiologic energy expenditure index will be calculated during the six-minute walk test.

When we examine the literature, there are many separate studies on the alignment of the pelvis after stroke, weight transfer symmetry, postural control and energy consumption of individuals with stroke. However, there is a lack of studies on spinal alignment in stroke patients in general. Therefore, the aim of this study was to investigate the relationship between spinal alignment, posture and weight transfer symmetry with balance, physical performance and energy expenditure in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 18-75 years diagnosed with stroke
* Volunteering to participate in the study
* Diagnosis of hemorrhagic or ischemic stroke,
* No collaboration and communication problems
* Can walk with assistive device or independently

Exclusion Criteria:

* Have another neurological, cardiopulmonary or orthopedic problem other than stroke that may affect functionality, ambulation and balance
* Patients who refused to participate in the study and did not give written consent.
* Cooperation and communication problems were determined as

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals aged 18-75 years with ischemic or hemorrhagic stroke who applied to Kırıkkale University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation will be included in our study
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2025-06-18 (Estimated); Study Completion 2025-07-05 (Estimated)

PRIMARY OUTCOMES:
Use of Spinal Mouse | day 1
  The SM device is started at the 7th cervical vertebra and advanced to the anal line. During the measurement, the mouse is lowered from the skin surface at a constant speed from top to bottom at the midpoint of the processus spinosus. Individuals are asked to assume the upright, maximal flexion, maximal extension positions in sequence.
  The relevant parameters in each position are thoracic curvature angle, lumbar curvature angle, sacrum-hip angle, tilt angle, mobility assessment (from extension to flexion position). The data transferred by the SM device to the computer via Bluetooth is analyzed and the angular deviation between each vertebra is calculated by the SM software as an angle value. The raw data of the wireless and handheld mouse is transferred to the computer via bluetooth and the data is analyzed by the SM software.
Postural Symmetry Index | day 1
  A form of measurement in which two scales are used to calculate the weight transferred to the intact and paralyzed limb. The values obtained as a result of the test are calculated with the following formulas. In this index, percentages close to 0 define equal symmetry and good postural control while standing, while higher percentages define asymmetry and poor postural control. Postural Symmetry (%) = Weight on Paralytic Side / Body Weight - 0.5| x 100 Weight Transfer Symmetry = Weight on Intact Side - Weight on Paralytic Side (%) Total Body Weight.
The Postural Assessment Scale (PASS) | day 1
  The PASS contains 12 items that measure a person's balance performance in situations of varying difficulty, such as lying, sitting, standing or changing standing position. The scale is administered under two main headings: during posture maintenance and posture change. Sitting without support, standing with support, standing without support, standing on paretic and nonparetic legs are the balance assessments under the heading of maintaining posture. Lateral rotation from supine to paretic and nonparetic side, lateral rotation from supine to sitting, from sitting to supine, from sitting to supine, from sitting to supine, from sitting to standing, from standing to sitting, and picking up a pen on the floor while standing are balance assessments under the heading of posture change. The scale is evaluated between 0-36. The feasibility of the movement is tested between 0-3; "0" is the lowest value; "3" is the highest value
MINI-BEST TEST | day 1
  Mini-BEST Test will be used to determine balance level. It consists of 4 sub-parameters including preparatory movement, reactive postural control, sensory orientation, dynamic walking and a total of 14 items. It is a test that is evaluated over a total of 28 points and requires an average of 10-15 minutes. High score indicates high function
Functional reach test (FRT) | day 1
  It is used to measure both the individual's functional balance and the amount of dynamic reaching. Patients will first be asked to extend their arm straight forward and the distance they reach will be recorded. They will then be asked to reach as far as they can reach forward without lifting their heels off the floor. The maximum value at which he/she can reach and return to his/her original position without losing his/her balance will be measured. Repeating 3 times, these three values will be averaged
Timed Up and Go Test (TUG) | day 1
  The timed stand and walk test (STWT) is used to assess timed performance. In the application, the individual first gets up from the chair, walks 3 meters, then walks back to the same chair and sits down again. The patient's time to complete the test is measured with a stopwatch. Measuring the time taken during this performance is used to determine the functional mobility of the person. Accordingly, completing the task in ≤ 10 seconds indicates that functional mobility is normal, completing the task in 10-20 seconds indicates that mobility is good, the person can walk with or without a device, can go out alone, completing the task in 20-30 seconds indicates that there is a serious problem with mobility and that the person performs mobility using an assistive device.
6 Minute Walk Test(6MWT) | day 1
  6 Minute Walk Test (6MWT): Physiological expenditure index (PEI) will be calculated to evaluate the energy expenditure and walking effort of individuals during the test. During the test, individuals will be asked to walk as fast as possible in a 30-meter straight corridor. Individuals will be told that if they feel tired or breathless during the test, they can rest or stop the test. Standard words of encouragement are used during the test. At the end of the test, the 6MWT distance is recorded in meters. Using age and gender, 6MWT expected values and 6MWT distance (% 6MWT) values expressed as a percentage of the expected values (6MWT distance * Body weight (kg)) are calculated. A 6MWT distance of less than 82% indicates a reduced functional capacity
The Five Times Sit to Stand Test (5xSTS) | day 1
  For the test, the individual is asked to sit on a chair with a height of 43.18 (12 inches) cm with the back straight, feet in contact with the floor and arms crossed on the chest. The individual is asked to sit on and stand up from the chair 1 time for a trial. After the trial performance, he/she is instructed to sit on the chair and stand up as quickly as possible and without stopping, and the elapsed time at the end of the fifth repetition is recorded. Validity and reliability studies were conducted in individuals with stroke 20-29 yrs ⇒ 6.0±1.4 sec 30-39 yrs ⇒ 6.1±1.4 sec 40-49 yrs ⇒ 7.6±1.8 sec 50-59 yrs ⇒ 7.7±2.6 sec 60-69 yrs ⇒ 8.4±0.0 sec (male), 12.7±1.8 sec (female) 70-79 yrs ⇒ 11.6±3.4 sec (male), 13.0±4.8 sec (female) 80-89 yrs ⇒ 16.7±4.5 sec (male), 17.2±5.5 sec (female) 90+ yrs ⇒ 19.5±2.3 sec (male), 22.9±9.6 sec (female)
Measurement of the craniovertebral angle | day 1
  Measurement of the craniovertebral angle; the patient is asked to find the most natural position by flexion and extension of the head in the standing position and a photograph is taken with a digital camera from a distance of 1.5 m to the shoulder level of the patient and this process is repeated 3 times. The images obtained are then digitally calculated with the help of an appropriate program.

CONTACTS AND LOCATIONS:
Overall Officials: Saniye Arslan, Assoc.Prof., Principal Investigator — Kırıkkale University; Serhat Ceylan, PT, MSc., Principal Investigator — Kırıkkale University
Locations (1):
- Kırıkkale University, Kırıkkale, Turkey (Türkiye)